CLINICAL TRIAL: NCT04331028
Title: Effect of Shock-wave Therapy on the Resorption and Bone Formation in Maxillary Postextraction Sockets
Acronym: Shockwave
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sctrict inclusion and exclusion criteria made the study unfeasible. No patients were enrolled.
Sponsor: Rui Figueiredo (Other)
Collaborators: MTS Europe GmbH (sponsor) (Unknown)
Responsible Party: Sponsor-Investigator, Rui Figueiredo, Associate Professor; IDIBELL researcher, University of Barcelona
Organization: University of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 496/14/EC; 496/14/EC (Other: AEMPS); 15/2013 (Other: CEIC Hospital Odontologic)
Record Dates: First submitted 2014-12-11; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Loss of Teeth Due to Extraction; Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shockwave therapy (Experimental): After dental extraction, a shockwave therapy will be applied to the area.
  Interventions: Device: Shockwave therapy
- Control (No Intervention): After dental extraction, no treatment will be applied

INTERVENTIONS:
Device: Shockwave therapy — A shockwave therapy device will be applied in the alveolar socket area of a maxillary tooth, 2 weeks after tooth extraction was performed.
  Arms: Shockwave therapy

SUMMARY:
The extracorporeal shock wave therapy (ESWT) has shown good results in bones and soft tissues of the lower and upper extremities such as: pseudoarthrosis, promoting bone formation of delayed or nonunion fractures, tendinopathies, fascitis and even in vascular pathologies.

The investigators main hypothesis is that the application of extracorporeal shock wave therapy (ESWT) in the residual alveolar bone after an extraction of an anterior upper maxillary tooth should prevent further residual alveolar bone resorption and will enhance vital bone formation.

The investigators null hypothesis is that applying extracorporeal shock wave therapy (ESWT) in the residual alveolar bone after an extraction of an anterior upper maxillary tooth has no influence in the alveolar bone remodeling process.

Therefore, the investigators main objective is to evaluate the efficacy of the ESWT in the prevention of alveolar bone resorption after an extraction with a volumetric exam through computer tomographies (CT) analysis. The investigators secondary objective is to determine the effect of ESWT in the internal bone healing process of these postextraction alveolar sockets, measuring the bone density in the CT (Hounsfield units) and the histomorphometric exam.

Methodology: randomized and open clinical trial with 20 patients (10 per group: with or without ESWT treatment) that comply the inclusion and exclusion criteria. In the first appointment the tooth extraction will be performed, while in the second visit (two weeks later), CT scan will be made to all patients and ESWT will be applied in the experimental group. Finally, in the third visit (ten weeks later), a new CT scan will be done and an implant will be placed in the zone taking previously a bone sample with a trephine bur.

The expected results are an improvement in the quantity and quality of the alveolar bone before the implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 - 65 years old.
* Non-smoking patients.
* Patients committed to rehabilitate the extraction socket with an implant.
* Lack of pathology in the surrounding area.
* Cooperative patients with serious commitment to follow the investigator's postoperative visits, who must sign the informed consent.
* Patients that need a conventional anterior maxillary single tooth extraction.

Exclusion Criteria:

* Systemic illnesses (ASA III or above) that could contraindicate a surgical intervention or modify the wound healing.
* Patients with cardiopathies.
* Patients taking hormones, calcium or oral or endovenous bisphosphonates.
* Patients with uncontrolled periodontitis / periimplantitis.
* Smokers.
* Patients with implant/s in the upper maxilla.
* Surgical extractions that require rising a flap or ostectomy.
* Bone defects larger of 2 mms in alveolar sockets due to cortical bone defect or resorption, fenestrations or/and dehiscences.
* Guided bone regeneration need.
* Periapical radiolucency larger than 2-3 mms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Bone volume | 10 weeks
  Measured in Cone Beam Computer Tomography
Histomorphometry | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rui Rui, DDS, MS, PhD, Principal Investigator — University of Barcelona
Locations (1):
- Hospital Odontologic, L'Hospitalet de Llobregat, Barcelona, Spain